CLINICAL TRIAL: NCT01858103
Title: A Multicenter, Open-label BMN 110 US Expanded Access Program (BMN 110 US EAP) to Provide BMN 110 to Patients Diagnosed With MPS IVA
Brief Title: BMN 110 US Expanded Access Program
Status: Approved for marketing | Type: Expanded Access
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 110-503
Record Dates: First submitted 2013-05-15; First posted 2013-05-21 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Mucopolysaccharidosis IVA; Morquio A Syndrome; MPS IVA
Keywords: Mucopolysaccharidosis IVA Type A; MPS IVA Type A; Mucopolysaccharidosis IVA; MPS IVA; Morquio A Syndrome; Lysosomal Storage Disorder; LSD; N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate
MeSH Terms: conditions — Mucopolysaccharidosis IV; Lysosomal Storage Diseases | interventions — GALNS protein, human

INTERVENTIONS:
Drug: BMN 110

SUMMARY:
The Expanded Access Program (EAP) is an open-label, multicenter program to:

1. Provide patients who have been diagnosed with Mucopolysaccharidosis IVA (MPS IVA) access to BMN 110 until commercial product is available
2. Collect additional information on the safety and tolerability of BMN 110 administration in patients with MPS IVA

Patients enrolled in the EAP will receive 2.0 mg/kg intravenous infusions of BMN 110 every week during the program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MPS IVA as confirmed by either N-acetylgalactosamine-6-sulfatase (GALNS) enzymatic test (GALNS activity in affected range, beta-galactosidase and a second lysosomal sulfatase activity within normal range) or molecular diagnostic test (two mutations in GALNS identified that have previously been associated with an enzyme defect).
* Willing and able to provide written, signed informed consent, or in the case of patients under the age of 18, provide written assent (as required by the IRB) and written informed consent by a legally authorized representative after the nature of the program has been explained, and prior to any program assessments or evaluations.
* Sexually active patients must be willing to use an acceptable method of contraception while participating in the program.
* Females of childbearing potential must have a negative pregnancy test at Baseline and be willing to have additional pregnancy tests during the program.
* Willing and able to comply with all program procedures.

Exclusion Criteria:

* Pregnant or breastfeeding at Baseline or planning to become pregnant (self or partner) at any time during the program. Patients who become pregnant during the program will be discontinued from the program.
* Currently enrolled in an ongoing clinical study of BMN 110.
* Discontinued from a BMN 110 clinical study secondary to a safety-related event.
* Use of any investigational product (other than BMN 110 in a clinical study) or investigational medical device within 30 days prior to Baseline, or requirement for any investigational agent prior to completion of all scheduled program assessments.
* Not a current US resident or expecting to have travel plans outside the US during the planned period of participation in the Expanded Access Program (EAP) that may interfere with dosing regimen, scheduled program visits and safety monitoring.
* Any condition that, in the view of the Investigator or sponsor, places the patient at high risk of poor treatment compliance or of not completing the EAP.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (25):
- United States (24):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Oakland, California
  - Orange, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Hollywood, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Minneapolis, Minnesota
  - Paterson, New Jersey
  - Manhasset, New York
  - New York, New York
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Tacoma, Washington
- Santurce, Puerto Rico